CLINICAL TRIAL: NCT05765708
Title: The Effect of Motor Imagery and Action Observation on Motor Skill Acquisition in Healthy Adults
Brief Title: The Effect of Motor Imagery and Action Observation on Motor Skill Acquisition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istinye University (Other); Ufuk University (Other)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Primary Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstanbulMU87
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motor imagery group (Experimental): Motor imagery group. Only motor imagery intervention will be applied to participants.
  Interventions: Other: Motor Imagery
- Action Observation Group (Experimental): Action Observation Group. Only action observation intervention will be applied to participants
  Interventions: Diagnostic Test: Action Observation
- Action Observation + Motor imagery Group (Experimental): Action Observation + Motor imagery Group. Both action observation and motor imagery interventions will be applied for 5 minutes each.
  Interventions: Other: Motor Imagery; Diagnostic Test: Action Observation
- Control (No Intervention)

INTERVENTIONS:
Other: Motor Imagery — Motor imagery is the mental execution of a movement without any overt movement or without any peripheral (muscle) activation. It has been shown that motor imagery leads to the activation of the same brain areas as an actual movement. Therefore, it is used to acquire new motor skills. Action Observation (AO) involves the dynamic process of observing purposeful actions with the intention of imitating and then practicing those actions.
  Arms: Action Observation + Motor imagery Group; Motor imagery group
Diagnostic Test: Action Observation — Action Observation (AO) involves the dynamic process of observing purposeful actions with the intention of imitating and then practicing those actions.
  Other Names: Movement Observation
  Arms: Action Observation + Motor imagery Group; Action Observation Group

SUMMARY:
The aim of this study is to investigate the effects of Motor Imagery and Action Observation on Motor Skill Acquisition in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Right hand dominance

Exclusion Criteria:

* Individuals with neurological, orthopedic, or rheumatological disease (for example: stroke, essential tremor, tennis player, trigger finger, rheumatoid arthritis, etc.)
* Severe cognitive problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Finger Tapping Task | 5 minutes
  The finger tapping task is a motor sequence learning task in which participants are asked to tap with their non-dominant hand a 5-digits sequence (for example 4-1-3-2-4 or 2-4-13-2), as rapidly and accurately as possible, using the numeric key-buttons of a computer keyboard or a response box.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire-3 | 15 minutes
  The Movement Imagery Questionnaire-3 is the most recent version of the Movement Imagery Questionnaire and the Movement Imagery Questionnaire-Revised. It is a 12-item questionnaire to assess individual's ability to image four movements using:
  Internal visual imagery External visual imagery Kinesthetic imagery. A 7 point scale used to score each item and the higher score indicates higher ability to perform motor imagery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No